CLINICAL TRIAL: NCT07023159
Title: Predicting Clinical Factors and Laboratory Parameters Associated With Short-Term Survival in Out-of-Hospital Cardiac Arrest
Brief Title: Predicting 28-Day Survival in OHCA Patients
Acronym: OHCAstd
Status: Completed | Type: Observational
Sponsor: Haseki Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Adem Az, Principal Investigator, Haseki Training and Research Hospital
Other Study IDs: 01-2023
Record Dates: First submitted 2025-05-26; First posted 2025-06-15 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Out of Hospital Cardiac Arrest; Cardiac Arrest (CA)
Keywords: OHCA; short-term survival; endotracheal intubation; cardiopulmonary resuscitation; neurological outcomes
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest; Heart Arrest | interventions — Demography; Comorbidity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Survivors: Survivors were defined as the patient being alive at 28 days following the cardiac arrest event.
  Interventions: Other: Demographics; Other: Comorbidities; Other: Prehospital Variables; Diagnostic Test: Hematological Parameters; Diagnostic Test: Biochemical Parameters; Diagnostic Test: Arterial Blood Gas Parameters
- Non-survivors: Non-survivors had passed away within 28 days following the cardiac arrest event.
  Interventions: Other: Demographics; Other: Comorbidities; Other: Prehospital Variables; Diagnostic Test: Hematological Parameters; Diagnostic Test: Biochemical Parameters; Diagnostic Test: Arterial Blood Gas Parameters

INTERVENTIONS:
Other: Demographics — The demographic profile of each patient was documented, including age and sex, to examine potential associations with survival and neurological outcomes.
Other: Comorbidities — Data on pre-existing chronic conditions were recorded, such as hypertension, diabetes mellitus, coronary artery disease, chronic kidney disease, and malignancy, in order to assess their potential impact on prognosis following OHCA.
Other: Prehospital Variables — Several prehospital factors were evaluated, including whether the cardiac arrest was witnessed, whether bystander CPR was performed, the time from collapse to the initiation of CPR, and the time from collapse to EMS arrival. Additionally, the durations of no-flow (i.e., time without any CPR) and low-flow (i.e., time with CPR but without ROSC) were noted. The initial cardiac rhythm was categorized as ventricular fibrillation or pulseless ventricular tachycardia (VF/pVT), asystole, or pulseless electrical activity (PEA). Airway management methods used in the field were documented and classified as bag-valve-mask (BVM), supraglottic airway devices (SGAs), or endotracheal intubation (ETI). Other recorded interventions included prehospital defibrillation, administration of epinephrine (including total dosage), and use of mechanical chest compression devices. Whether ROSC was achieved prior to arrival at the emergency department was also noted.
Diagnostic Test: Hematological Parameters — These included white blood cell count (WBC), hemoglobin level, platelet count, mean platelet volume (MPV), and differential counts such as neutrophils, monocytes, and eosinophils.
Diagnostic Test: Biochemical Parameters — Measurements included creatinine, urea, lactate dehydrogenase (LDH), aspartate aminotransferase (AST), alanine aminotransferase (ALT), sodium, potassium, chloride, calcium, and troponin-I levels.
Diagnostic Test: Arterial Blood Gas Parameters — The primary clinical outcomes recorded for each patient included return of spontaneous circulation (ROSC), 28-day survival or mortality, and neurological status, which was later assessed using the Cerebral Performance Category (CPC) scale.

SUMMARY:
This prospective study aimed to identify clinical and laboratory predictors of return of spontaneous circulation (ROSC), 28-day survival, and favorable neurological outcomes in adult patients experiencing out-of-hospital cardiac arrest (OHCA) and brought to the emergency department (ED) by emergency medical services (EMS). Specifically, the prognostic value of hematologic, biochemical, and blood gas parameters on admission was assessed for ROSC, 28-day survival, and favorable neurological recovery. Additionally, the study investigated the influence of key patient-centered and prehospital variables, including demographic features, initial cardiac rhythm, and the timeliness and type of cardiopulmonary resuscitation (CPR), defibrillation, and airway interventions, on overall survival and neurological status.

DETAILED DESCRIPTION:
This prospective, observational, and cross-sectional study was conducted in the ED of a tertiary urban hospital between May 2023 and May 2024. Adult patients (aged ≥18 years) who experienced OHCA and received attempted resuscitation by EMS personnel were screened for eligibility. All patients received advanced cardiac life support (ACLS) in accordance with the 2021 European Resuscitation Council (ERC) and 2020 American Heart Association (AHA) guidelines.

Patients were initially categorized into survivors and non-survivors based on ROSC and 28-day survival status. Furthermore, 28-day survivors were stratified into two subgroups based on their neurological status using the Cerebral Performance Category (CPC) score. Favorable neurological outcome was defined as CPC 1-2 (good to moderate cerebral performance with independence), while CPC 3-5 (severe disability, coma, or death) constituted unfavorable outcome.

Prior to the initiation of the study, a standardized and pre-piloted data collection form was developed based on current literature to ensure consistency and reproducibility. During the study period, patient data were initially recorded by board-certified emergency medicine specialists who were on duty in the ED at the time of each patient's arrival. These attending physicians were directly responsible for patient management and completed the data forms either during the resuscitation process or immediately thereafter. All physicians involved in data entry were blinded to the study hypothesis. Subsequently, all collected data were extracted, cross-checked, and verified for accuracy and completeness by an emergency medicine specialist with eight years of clinical experience, who was also blinded to the study hypothesis.

Patient data were obtained from multiple sources, including hospital's automated systems and ED's archives, prehospital EMS reports, and the national digital healthcare database of Türkiye (e-Nabız), which was used to verify survival status and neurological outcomes at 28 days.

Collected data includes, demographics (age, sex), comorbidities (hypertension, diabetes mellitus, coronary artery disease, chronic kidney disease, or malignancy), and prehospital variables such as whether the cardiac arrest was witnessed, whether bystander CPR was performed, the time from collapse to the initiation of CPR, the time from collapse to EMS arrival, the durations of no-flow (time without CPR) and low-flow (time with CPR but no ROSC), and the initial cardiac rhythm, categorized as ventricular fibrillation or pulseless ventricular tachycardia (VF/pVT), asystole, or pulseless electrical activity (PEA). The airway management method used by EMS was also recorded, including BVM, SGD, or ETI. Other recorded interventions included prehospital defibrillation, epinephrine administration (including total dose), and the use of mechanical chest compression devices. Whether ROSC was achieved in the field prior to ED arrival was also documented.

On arrival to the ED, clinical examination findings included the patient's body temperature, the Glasgow Coma Score (if measurable), the presence or absence of pupillary light reflex, and the requirement for vasopressor support within the first hour.

Laboratory data obtained upon admission included hematological parameters such as white blood cell count (WBC), hemoglobin level, platelet count, mean platelet volume (MPV), neutrophil count, monocyte count, and eosinophil count. Biochemical measurements included creatinine, urea, lactate dehydrogenase (LDH), aspartate aminotransferase (AST), alanine aminotransferase (ALT), sodium, potassium, chloride, calcium, and troponin-I levels. Arterial blood gas analysis results included pH, partial pressure of carbon dioxide (pCO₂), bicarbonate, lactate concentration, carboxyhemoglobin percentage, and methemoglobin percentage.

Clinical outcomes, including ROSC, 28-day survival or mortality, and neurological status, were also recorded.

Patients' demographics, initial rhythm, prehospital intubation status, and hematological, biochemical, and blood gas parameters on admission were compared to identify factors associated with 28-day survival and neurological status between the groups. Independent predictors of survival were determined via multivariate logistic regression analysis of variables that significantly differed between survivors and non-survivors.

ELIGIBILITY:
Inclusion Criteria:

- This study included 420 adult patients (aged ≥18 years) who were brought to our hospital's ED due to OHCA and who had initiated attempted resuscitation by EMS were initially screened for inclusion between May 2023 and May 2024.

Exclusion Criteria:

* Patients aged < 18 years
* Patients with in-hospital cardiac arrest
* Patients who have suffered cardiac arrest due to major trauma, drowning, drug overdose, or known terminal illness
* Patients with active hematologic malignancy
* Patients with incomplete data regarding primary outcomes or admission laboratory tests

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study included 420 adult patients (aged ≥18 years) who were brought to our hospital's ED due to OHCA and who had initiated attempted resuscitation by EMS were initially screened for inclusion between May 2023 and May 2024.
Sampling Method: Probability Sample
Enrollment: 327 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Return of Spontaneous Circulation (ROSC) | Assessed within the first 20 minutes after emergency department admission.
  ROSC was defined as the return of sustained spontaneous perfusing rhythm lasting at least 20 minutes without the need for external chest compressions.
Number of Participants Alive at Day 28 | Assessed within the first 20 minutes after emergency department admission.
  Survival was assessed as the patient being alive at 28 days following the cardiac arrest event.
Number of Participants with Favorable Neurological Outcome (CPC 1-2) at Day 28 | Assessed within the first 20 minutes after emergency department admission.
  Neurological outcome was determined using the Cerebral Performance Category (CPC) scale, with a CPC score of 1 or 2 representing a favorable neurological outcome, and scores from 3 to 5 considered unfavorable, reflecting severe neurological disability, coma, or death.

SECONDARY OUTCOMES:
Comparison of 28-Day Survival Rates Between Participants Who Underwent Prehospital Endotracheal Intubation and Those Who Did Not | Assessed within the first 20 minutes after emergency department admission.
  The investigators evaluate the impact of prehospital endotracheal intubation (ETI) on 28-day survival status. Survival was defined as being alive 28 days after the cardiac arrest event. Participants will be categorized into two groups based on whether or not they received ETI in the prehospital setting.
Comparison of Favorable Neurological Outcome Rates at Day 28 Between Participants Who Underwent Prehospital Endotracheal Intubation and Those Who Did Not | Assessed within the first 20 minutes after emergency department admission.
  The investigators evaluate the impact of prehospital endotracheal intubation (ETI) on neurological outcomes at Day 28 following cardiac arrest. Neurological status will be assessed using the Cerebral Performance Category (CPC) scale. A CPC score of 1 or 2 will be considered a favorable neurological outcome. Participants will be categorized into two groups based on whether or not they received ETI in the prehospital setting.
Correlation Between Admission Serum Lactate Level and 28-Day Survival | Assessed within the first 20 minutes after emergency department admission.
  The investigators evaluate the correlation between serum lactate level at emergency department admission and 28-day survival status following out-of-hospital cardiac arrest. Lactate will be measured in mmol/L using a standard arterial blood gas analyzer.

CONTACTS AND LOCATIONS:
Overall Officials: Adem Az, Principal Investigator — Haseki Training and Research Hospital
Locations (1):
- Haseki Training and Research Hospital, Istanbul, Sultangazi, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Stored in non-publicly avaliable Avaliable on request

REFERENCES:
- [Background] Jabre P, Penaloza A, Pinero D, Duchateau FX, Borron SW, Javaudin F, Richard O, de Longueville D, Bouilleau G, Devaud ML, Heidet M, Lejeune C, Fauroux S, Greingor JL, Manara A, Hubert JC, Guihard B, Vermylen O, Lievens P, Auffret Y, Maisondieu C, Huet S, Claessens B, Lapostolle F, Javaud N, Reuter PG, Baker E, Vicaut E, Adnet F. Effect of Bag-Mask Ventilation vs Endotracheal Intubation During Cardiopulmonary Resuscitation on Neurological Outcome After Out-of-Hospital Cardiorespiratory Arrest: A Randomized Clinical Trial. JAMA. 2018 Feb 27;319(8):779-787. doi: 10.1001/jama.2018.0156. PMID 29486039
- [Background] Wang HE, Schmicker RH, Daya MR, Stephens SW, Idris AH, Carlson JN, Colella MR, Herren H, Hansen M, Richmond NJ, Puyana JCJ, Aufderheide TP, Gray RE, Gray PC, Verkest M, Owens PC, Brienza AM, Sternig KJ, May SJ, Sopko GR, Weisfeldt ML, Nichol G. Effect of a Strategy of Initial Laryngeal Tube Insertion vs Endotracheal Intubation on 72-Hour Survival in Adults With Out-of-Hospital Cardiac Arrest: A Randomized Clinical Trial. JAMA. 2018 Aug 28;320(8):769-778. doi: 10.1001/jama.2018.7044. PMID 30167699
- [Background] Strnad M, Borovnik Lesjak V, Jerot P, Esih M. Prehospital Predictors of Survival in Patients with Out-of-Hospital Cardiac Arrest. Medicina (Kaunas). 2023 Sep 26;59(10):1717. doi: 10.3390/medicina59101717. PMID 37893434
- [Background] Brooks SC, Clegg GR, Bray J, Deakin CD, Perkins GD, Ringh M, Smith CM, Link MS, Merchant RM, Pezo-Morales J, Parr M, Morrison LJ, Wang TL, Koster RW, Ong MEH; International Liaison Committee on Resuscitation. Optimizing Outcomes After Out-of-Hospital Cardiac Arrest With Innovative Approaches to Public-Access Defibrillation: A Scientific Statement From the International Liaison Committee on Resuscitation. Circulation. 2022 Mar 29;145(13):e776-e801. doi: 10.1161/CIR.0000000000001013. Epub 2022 Feb 15. PMID 35164535
- [Background] Soholm H, Wachtell K, Nielsen SL, Bro-Jeppesen J, Pedersen F, Wanscher M, Boesgaard S, Moller JE, Hassager C, Kjaergaard J. Tertiary centres have improved survival compared to other hospitals in the Copenhagen area after out-of-hospital cardiac arrest. Resuscitation. 2013 Feb;84(2):162-7. doi: 10.1016/j.resuscitation.2012.06.029. Epub 2012 Jul 13. PMID 22796541
- [Background] Bro-Jeppesen J, Kjaergaard J, Horsted TI, Wanscher MC, Nielsen SL, Rasmussen LS, Hassager C. The impact of therapeutic hypothermia on neurological function and quality of life after cardiac arrest. Resuscitation. 2009 Feb;80(2):171-6. doi: 10.1016/j.resuscitation.2008.09.009. Epub 2008 Dec 25. PMID 19111378